CLINICAL TRIAL: NCT00633152
Title: A Phase 2, Multicenter, Randomized, Open-label, Comparative Study to Evaluate the Efficacy and Safety of Intramuscular Ceftaroline Versus Intravenous Linezolid in Adult Subjects With Complicated Skin and Skin Structure Infections
Brief Title: Efficacy and Safety of Ceftaroline Versus Linezolid in Subjects With Complicated Skin and Skin Structure Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P903-19
Record Dates: First submitted 2008-03-03; First posted 2008-03-11 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Bacterial Infection
Keywords: complicated skin and skin structure infections; linezolid; ceftaroline; clinical response; microbiological response; Cellulitis; Abscess; Wound infection; Deeper soft tissue; Significant surgical intervention; Gram-positive bacterial infection; Gram-negative bacterial infection; bacterial infection; cephalosporin; broad-spectrum activity
MeSH Terms: conditions — Bacterial Infections; Cellulitis; Abscess; Wound Infection; Gram-Positive Bacterial Infections; Gram-Negative Bacterial Infections | interventions — Ceftaroline; Injections; Linezolid; Aztreonam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceftaroline (Experimental): Intramuscular every 12 hours
  Interventions: Drug: ceftaroline
- linezolid plus optional aztreonam (Active Comparator): Intravenous every 12 hours
  Interventions: Drug: linezolid; Drug: Aztreonam

INTERVENTIONS:
Drug: ceftaroline — 600 mg injected every 12 hours for at least 5 but not more than 14 days
  Other Names: ceftaroline fosamil; ceftaroline for injection
  Arms: Ceftaroline
Drug: linezolid — 600 mg parenteral infused over 60 minutes for a minimum of 5 days and a maximum of 14 days
  Other Names: Zyvox; Zyvoxid; CAS number 165800-03-3
  Arms: linezolid plus optional aztreonam
Drug: Aztreonam — 1000 mg infused over 60 minutes every 24 hours may be started with linezolid or added later (up to 72 hours after the first dose of linezolid) for subjects with a gram-negative infection indicated.
  Arms: linezolid plus optional aztreonam

SUMMARY:
The purpose of this study is to determine whether ceftaroline is effective and safe in the treatment of complicated skin and skin structure infections in adults.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether ceftaroline is effective and safe in the treatment of complicated skin and skin structure infections in adults. The primary focus is bacterial infection.

ELIGIBILITY:
Inclusion Criteria:

* Complicated skin and skin structure infection (cSSSI)
* Require initial hospitalization, or treatment in an emergency room or urgent care setting

Exclusion Criteria:

* Hypersensitivity or allergic reaction to any ß-lactam, ceftaroline, linezolid, aztreonam, or to their components
* Concomitant use of adrenergic or serotonergic agent
* Uncomplicated skin and skin structure infection
* Concomitant therapy with any drug known to exhibit a contraindicated drug-drug interaction
* More than 24 hours of treatment with an antimicrobial within 96 hours before randomization
* Known or suspected endocarditis, osteomyelitis, or septic arthritis
* Severely impaired renal function
* Evidence of significant hepatic, hematologic, or immunologic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor Cerexa, Study Director — Forest Laboratories
Locations (13):
- United States (13):
  - Investigational Site, Buena Park, California
  - Investigational Site, Long Beach, California
  - Investigational Site, Los Angeles, California
  - Investigational Site, Rolling Hills Estate, California
  - Investigational Site, San Diego, California
  - Investigational Site, Atlantis, Florida
  - Investigational Site, Columbus, Georgia
  - Investigational Site, Savannah, Georgia
  - Investigational Site, Minneapolis, Minnesota
  - Investigational Site, Butte, Montana
  - Investigational Site, Somers Point, New Jersey
  - Investigational Site, Columbus, Ohio
  - Investigational Site, Toledo, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve (12) study centers in the U.S. participated in this open label trial.
Groups:
- Linezolid: Intravenous Linezolid every 12 hours (with or without Aztreonam)
Period: Overall Study
Arm/Group | Ceftaroline | Linezolid
Started | 103 | 47
MITT and Safety Population | 98 | 45
Clinically Evaluable Population | 86 | 39
Completed | 89 | 41
Not Completed | 14 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Randomized, did not receive study drug | 5 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 4 | 1
Not completed — Miscellaneous Other | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftaroline | Linezolid | Total
Number analyzed (Participants) | 103 | 47 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (12.83) | 39.9 (14.58) | 39.7 (13.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 18 | 51
  Male | 70 | 29 | 99
Region of Enrollment [Number; unit: participants]
  United States | 103 | 47 | 150

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response at the Test of Cure (TOC) Visit in the Modified Intent-to-treat (MITT) Population
Description: The coprimary efficacy outcome measures were the per-subject clinical cure rate at the Test of Cure (TOC) Visit in the Clinically Evaluable (CE) and (Modified-Intent-to-Treat) MITT Populations. Subjects were considered clinically cured at the Test of Cure (TOC) Visit if they had total resolution of all signs and symptoms of the baseline infection, or improvement of the infection to such an extent that no further antimicrobial therapy was necessary.
Time Frame: Test of Cure Visit (8 to 15 days after end of therapy)
Population: Modified-Intent-to-Treat (MITT) Population - Any randomized subjects that received any amount of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Ceftaroline: Ceftaroline was administered 600 mg as an Intramuscular injection every 12 hours
- Linezolid (With or Without Aztreonam): Linezolid was administered as 600 mg Intravenous infusions over 60 minutes every 12 hours
Arm/Group | Ceftaroline | Linezolid (With or Without Aztreonam)
Number analyzed (Participants) | 98 | 45
percentage of participants | 84.7 [76.0 to 91.2] | 88.9 [75.9 to 96.3]

2. Primary Outcome: Clinical Response at the Test-of-Cure (TOC) Visit in the Clinically Evaluable (CE) Population
Description: The coprimary efficacy outcome measures were the per-subject clinical cure rate at the TOC Visit in the CE and MITT Populations. Subjects were considered clinically cured at the TOC Visit if they had total resolution of all signs and symptoms of the baseline infection, or improvement of the infection to such an extent that no further antimicrobial therapy was necessary.
Time Frame: Test of Cure Visit (8 to 15 Days after end of therapy)
Population: The Clinically Evaluable (CE) Population included all subjects who satisfied key minimum protocol criteria
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Ceftaroline: Ceftaroline fosamil was administered 600mg IM every 12 hours
- Linezolid (With or Without Aztreonam): Linezolid was administered as 600 mg IV infusions over 60 minutes q12h
Arm/Group | Ceftaroline | Linezolid (With or Without Aztreonam)
Number analyzed (Participants) | 86 | 39
percentage of participants | 90.7 [82.5 to 95.9] | 97.4 [86.5 to 99.9]

3. Secondary Outcome: Clinical Cure Rate at the TOC Visit in the cMITT Population
Description: Evaluate per-subject the clinical response at the Test-of-Cure (TOC) Visit in the Clinical Modified Intent-to-treat (cMITT) Population.
Time Frame: TOC Visit (8 to 15 days after end of therapy)
Reporting Status: Not Posted

4. Secondary Outcome: Clinical Response at the End-of-Therapy (EOT) Visit in the MITT, cMITT and CE Populations.
Description: Evaluate per-subject the clinical response at the End-of-therapy (EOT) Visit in the MITT, cMITT and CE populations.
Time Frame: End-of-therapy (EOT) visit
Reporting Status: Not Posted

5. Secondary Outcome: The Microbiological Response at the TOC Visit in the mMITT and ME Populations.
Description: Evaluate per-subject the microbiological response at the TOC Visit in the Microbiological Modified Intent-to-treat (mMITT) and Microbiologically Evaluable (ME) populations.
Time Frame: TOC Visit (8 to 15 days after end of therapy)
Reporting Status: Not Posted

6. Secondary Outcome: Clinical and Microbiological Response by Pathogen at the TOC Visit in the mMITT and ME Populations
Description: Evaluate the clinical and microbiological response by pathogen at the TOC Visit in the mMITT and ME populations.
Time Frame: TOC Visit (8 to 15 days after end of therapy)
Reporting Status: Not Posted

7. Secondary Outcome: Clinical Relapse at the Late Follow-up Visit
Description: Evaluate Clinical relapse rate at Late Follow-up (LFU) (21 to 45 days after the final dose of study drug)in those subjects clinically cured at the TOC visit.
Time Frame: Late Follow-up (LFU) Visit (21 to 35 days after end of therapy)
Reporting Status: Not Posted

8. Secondary Outcome: The Microbiological Reinfection or Recurrence at the Late Follow-up (LFU) Visit
Description: Evaluate per-subject reinfection or recurrence rate at the LFU Visit in those subjects who had a favorable microbiological outcome (eradication or presumed eradication) at the TOC Visit.
Time Frame: LFU Visit (21 to 35 days after end of therapy)
Reporting Status: Not Posted

9. Secondary Outcome: The Safety of Ceftaroline Fosamil
Description: Evaluate safety of Ceftaroline fosamil IM in adults with complicated skin and skin structure infection (cSSSI)
Time Frame: First dose of study drug through LFU Visit or 30 days after the last dose of study drug
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Date of First Dose of study drug to the TOC visit (AEs) or LFU visit (SAEs).
Arm/Group | Ceftaroline | Linezolid
Serious Adverse Events (participants affected / at risk) | 4/98 | 0/45
Other Adverse Events (participants affected / at risk) | 35/98 | 15/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftaroline (N=98) | Linezolid (N=45)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Necrotizing fasciitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Postoperative wound infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftaroline (N=98) | Linezolid (N=45)
Nausea (Gastrointestinal disorders) | 12 (15) | 7 (11)
Headache (Nervous system disorders) | 10 (14) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 4 (4)
Injection site irritation (General disorders) | 6 (60) | 0 (0) — Administration site conditions
Somnolence (Nervous system disorders) | 6 (6) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dysgeusia (Nervous system disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No